CLINICAL TRIAL: NCT02231333
Title: A Randomized Controlled Trial to Study the Efficacy of S-adenosyl Methionine (SAMe) Versus Pentoxiphylline in Patients With Non-alcoholic Steatohepatitis With Fibrosis.
Brief Title: The Efficacy of S-adenosyl Methionine (SAMe) Versus Pentoxiphylline in Patients With Non-alcoholic Steatohepatitis With Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-NASH-01
Record Dates: First submitted 2014-08-30; First posted 2014-09-04 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-adenosylmethionine (SAMe) (Experimental)
  Interventions: Drug: S-adenosylmethionine (SAMe)
- pentoxiphylline (PTX) (Active Comparator)
  Interventions: Drug: pentoxiphylline (PTX)

INTERVENTIONS:
Drug: S-adenosylmethionine (SAMe)
  Arms: S-adenosylmethionine (SAMe)
Drug: pentoxiphylline (PTX)
  Arms: pentoxiphylline (PTX)

SUMMARY:
Nonalcoholic fatty liver disease is one the most commonly encountered conditions in a daily outpatient Hepatology clinic. Secondly our country is the diabetic capital of the world and so the incidence of NAFLD (Non Alcoholic Fatty Liver Disease) is expected to rise in the future. It is a spectrum of hepatic pathology, ranging from simple steatosis, steatohepatitis, to cirrhosis. Nonalcoholic steatohepatitis (NASH) is a more advanced form of disease where steatosis is accompanied by hepatocyte injury as well as infiltration of inflammatory cells. Approximately 10-20% of patients with NASH may progress to cirrhosis. NASH is felt to be a major etiology of cryptogenic cirrhosis. Around 6230 human studies out of which 49 RCTs have been done till date to define the appropriate treatment of nonalcoholic steatohepatitis. However, still a controversy and no recommended treatment available till date. Recently published PIVENS trial has shown that Vitamin E has proven benefit in NASH. Other trials have also shown that pentoxiphylline has shown benefit in the form of histological improvement and biochemical improvement in the form of liver enzymes. Role of SAMe has been studied in alcoholic liver disease and showed to improve in both biochemical and histological features. However the usefulness of SAMe in NAFLD is not known till now. Hence this study has been designed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Persistently abnormal ALT >1.2 times upper limit of normal
* Histological evidence of NASH (Non alcoholic Steatohepatitis) on liver biopsy. The minimal criteria for diagnosis of NASH included the presence of lobular inflammation and fibrosis up to stage 3 as per Burnt stating.

Exclusion Criteria:

* Alcohol intake of more than 40gm / week with features suggestive chronic liver disease .
* Other known cause of chronic liver disease like Hepatitis B,C, autoimmune liver disease, Wilson's disease, alpha 1 antitrypsin deficiency and hemochromatosis, primary biliary cirrhosis, PSC (Primary Sclerosis Cholangitis).
* Patient on Medication like estrogens, amiodarone, MTx, tamoxifen, ATT (Antitubercular Treatment)
* Pregnancy or lactation
* Hypersensitivity to methylxanthines (e.g., caffeine, theophylline,)
* Recent retinal/cerebral hemorrhage
* Acute myocardial infarction or severe cardiac arrhythmias.
* Impaired renal function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Biochemical improvement in the form of AST/ALT | 1 Years
Improvement in LSM (Liver Stiffness Measurement) & CAP (Controlled Attenuation Parameter) | 1 years

SECONDARY OUTCOMES:
Metabolic response in form of anthropometry. | 1 Years
  metabolic response in form of anthropometry (BMI, waist circumference).
Fasting lipid profiles | 1 Years
Reduction in uric acid levels | 1 Years
Reduction in pro- inflammatory cytokines | 1 Years
Histological outcome in the form of improvement or non- progression in hepatocyte injury and fibrosis. | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Devaraja R, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India